CLINICAL TRIAL: NCT01330823
Title: L-Carnitine in the Palliative Treatment of Advanced Pancreatic Cancer (CARPAN): a Prospective, Randomised, Placebo Controlled, Double Blinded, Multicentre Trial
Brief Title: L-CARnitine in the Palliative Treatment of Advanced PANcreatic Cancer (CARPAN)
Acronym: CARPAN
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: after interims analysis standard errors for inflammatory and nutritional markers varied widely, that the power calculation required unattainable goals
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Markus M Lerch, Professor of Medicine, Department of Medicine A
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CARPAN-01
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Pancreatic Carcinoma
Keywords: pancreatic carcinoma; L-Carnitine; quality of life; survival; malnutrition; cancer cachexia; fatigue
MeSH Terms: conditions — Pancreatic Neoplasms; Malnutrition; Fatigue | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-Carnitine (Active Comparator): L-Carnitine 4 g daily for Intervention
  Interventions: Dietary Supplement: L-Carnitine
- Placebo (Placebo Comparator): Placebo (tartaric acid)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Carnitine — L-Carnitine, 4g/day, orally (Juice)
  Arms: L-Carnitine
Dietary Supplement: Placebo — tartaric acid same dose like L-Carnitine as placebo
  Arms: Placebo

SUMMARY:
The study investigated the role of L-Carnitine supplementation on proinflammatory immune response, malnutrition, cancer cachexia and cancer related fatigue in advanced and inoperable pancreatic cancer, UICC Stage IV .

DETAILED DESCRIPTION:
Pancreatic cancer has the lowest 5-year survival rate of any cancer and ranks as the fourth leading cause of cancer death world wide. Several metabolic changes are present in the whole body in case of cancer so the investigators conducted a placebo controlled, double blinded, randomized, prospective and multicentre study to investigate, whether L-Carnitine supplementation may have an impact on malnutrition, cancer cachexia and cancer related fatigue in advanced pancreatic cancer.

Study drug: L-Carnitine 4g per day (vers) Placebo Study design: A multi-centre, double blind, and placebo-controlled, randomised, parallel group study

Patient population: Patients with advanced pancreatic carcinoma Number of patients: Total of 90 patients in two equal groups number of centres: 4 (Greifswald, Magdeburg, Berlin,Heidelberg,all Germany) Duration of dosing: 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* advanced pancreatic cancer (UICC Stage IV)
* Karnofsky Index larger than 60
* compliance
* consent to participate to the study

Exclusion Criteria:

* Child-Pugh classification of liver failure greater than Child B,
* a known second malignant tumor
* oral or parenteral supplementation with omega-3-fatty acids
* treatment with thalidomide or Infliximab
* mental or physical disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-06; Primary Completion 2009-10 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
TNF-alpha | 12 weeks
  Influence of L-Carnitine on proinflammatory cytokine TNF-alpha

SECONDARY OUTCOMES:
nutritional status | 12 weeks
  Bioelectrical impedance analysis (BIA) was performed,BCM / ECM index, phase angle, body fat was measured. Increase of body weight and body mass index and and also weight loss were investigated.
Quality of life | 12 weeks
  Quality of life was determined using the European EORTC QLQ-C30 form, along with an additional disease specific pancreatic cancer module PAN26 and also Brief Fatique Inventory (BFI).
survival | 1 year
  Survival time in days was calculated from time of diagnosis until death.
hospital stay | 1 year
  time of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Markus M. Lerch, Prof., Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald,Department of Medicine A, Greifswald, Germany

REFERENCES:
- See also: Related Info — http://www.pancreas.de